CLINICAL TRIAL: NCT06728462
Title: A Study Benchmarking FREEDOM Substudy to Evaluate the Effects of Amorphous Calcium Carbonate in Postmenopausal Women
Brief Title: A Study of Amorphous Calcium Carbonate in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universal Integrated Corp. (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UIC-DST-2024
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-12

CONDITIONS: Calcium; Osteoporosis; Bone Mineral Density; Bone Turnover Marker; Denosumab
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: External comparator arm study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A arm (Other): Subject who meet National Health Insurance (NHI) reimbursement criteria for use of denosumab
  Interventions: Dietary Supplement: Amorphous calcium carbonate
- B arm (Other): Subject who does not meet NHI reimbursement criteria for use of denosumab, or who is no willing to receive denosumab treatment during study period, even meet NHI reimbursement criteria
  Interventions: Dietary Supplement: Amorphous calcium carbonate

INTERVENTIONS:
Dietary Supplement: Amorphous calcium carbonate — The usual dose for oral use is 5 ACC tablets (equal to 1000 mg calcium element) daily given after meals.

SUMMARY:
Using the FREEDOM substudy as a benchmark, evaluate the effects of amorphous calcium carbonate (ACC) on bone mineral density (BMD) in postmenopausal women, both with and without the combination of Denosumab treatment.

DETAILED DESCRIPTION:
This is an open-label study to evaluate the effect of DensityTM, amorphous calcium carbonate (ACC), in postmenopausal women, compared to FREEDOM substudy.

Subjects with a BMD T-score between -4.0 to -2.5 will be invited to enroll into this study. After signed ICF, eligible subject who meet NHI reimbursement criteria for use of denosumab will be assigned to A arm, and subject who does not meet NHI reimbursement criteria for use of denosumab, or who is no willing to receive denosumab treatment during study period, even meet NHI reimbursement criteria will be assigned to B arm. A total of 205 subjects will be enrolled into this study, in which 142 subjects in A arm and 63 subjects in B arm.

In A arm, subject will receive 5 DensityTM tablets (equal to 1000 mg calcium element) daily with injections of 60 mg of ProliaTM (denosumab) every 6 months at study site, while in B arm, eligible subject will receive 5 DensityTM tablets (equal to 1000 mg calcium element) daily only. DensityTM tablets will be administered as follows: 5 tablets will be taken after meal. In addition, all subjects with a baseline 25-hydroxyvitamin D level of 12 to 20 ng/ml will be given 800 IU of vitamin D3 daily, while those with a baseline level above 20 ng/ml received 400 IU of vitamin D3, both administered after meal.

The study will consist of 7 clinical visits. Subjects will come to the clinics at Visit 1 (screening visit, Month -1), Visit 2 (regimen start, Day 0 in Month 0), and Visit 3 to 7 (follow-up visits, Month 1, 6, 12, 18, 24). BMD assessment and blood drawing will be performed before study medication administration and at Month 1, 6, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women who are 60 to 90 years of age.
2. With BMD T-score of lower than -2.5 at the lumbar spine or total hip and -4.0 or higher at both sites. Subject who also meet the following criteria:

   A arm:-Subject who meet National Health Insurance (NHI) reimbursement criteria for use of denosumab.

   B arm:-Subject who does not meet NHI reimbursement criteria for use of denosumab, or who is no willing to receive denosumab treatment during study period, even meet NHI reimbursement criteria.
3. Subject who are naïve to osteoporosis treatment or have received prior bisphosphonate treatment for less than 3 years and not within 12 months prior to screening visit.
4. A minimum of 2 evaluable lumbar vertebrae in the L1-L4 region and 1 evaluable hip (i.e., either the left or right side).
5. Willingness to limit additional Vitamin D3 intake to 400IU or 800IU per day during the study period.
6. Ability to complete the entire procedure and to comply with study instructions.
7. Will provide completed and signed written informed consent.

Exclusion Criteria:

1. Subjects who had conditions that influence bone metabolism (i.e., Paget's disease and osteomalacia).
2. Subject on other osteoporosis therapies, parathyroid hormone or its derivatives, corticosteroids, systemic hormone-replacement therapy, selective estrogen-receptor modulators, tibolone, calcitonin or calcitriol 6 weeks prior to screening visit.
3. Subjects had a serum 25-hydroxyvitamin D level of less than 12 ng/ml.
4. Subjects had a BMD T-score of less than -4.0 at the lumbar spine or total hip.
5. Subjects with any severe or more than two moderate vertebral fractures on spinal x-ray at screening visit.
6. Subject who plan to initiate a new bisphosphonate treatment during study period.
7. Known hypersensitivity to any component of the study drug product.
8. Participation in any other investigational study within 30 days prior to receiving study medication.
9. Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety.

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal Women
Enrollment: 205 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in LBMD | 2 years
  Percent change from baseline of bone mineral density (BMD) at the lumbar spine (L1, L2, L3, L4)

SECONDARY OUTCOMES:
Percentage change in BMD | 2 years
  Percent change from baseline of BMD at total hip, femoral neck, trochanter
Success rate in bone turnover markers (BTMs) | 2 years
  Percentage of Subjects with BTMs values, including P1NP and CTX, below the premenopausal reference interval at Month 0, 1, 6, 12, and 24. Premenopausal reference interval is defined as CTX values <0.20 ng/mL and P1NP values <17.4 ng/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No